CLINICAL TRIAL: NCT03933592
Title: Ultrasound Guided Serratus Plane Block Versus Thoracic Epidural for Post Thoracotomy Pain: A Prospective Randomized Controlled Study
Brief Title: Ultrasound Guided Serratus Plane Block Versus Thoracic Epidural for Post Thoracotomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Mamdouhmahmoud, Lecturer, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201617026
Record Dates: First submitted 2019-04-23; First posted 2019-05-01 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Ultrasound Guided Serratus Plane Block; Thoracic Epidural; Post Thoracotomy Pain
MeSH Terms: interventions — Tea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic epidural (Active Comparator): thoracic epidural inserted at low thoracic level in sitting position then test dose will be administered to detect any complications then a bolus of 10 ml of 0.25% levobupivacaine 30 mint before skin incision followed by an infusion of 5 ml/hour of 0.125% levobupivacaine after surgery.
  Interventions: Procedure: thoracic epidural
- Serratus plane block (Experimental): after induction of anesthesia and Patients will be placed in the lateral position with the diseased side up. A linear ultrasound transducer (10-12 MHz) will be placed over the mid-axillary region of the thoracic cage in a sagittal plane. The rib will be counted inferiorly and laterally until the fifth rib is identified in the mid-axillary line. The following muscles will be identified easily overlying the fifth rib: the latissimus dorsi (superficial and posterior), teres major (superior) and serratus muscle (deep and inferior). The needle (22- G, 50 - mm Touhy needle) will be introduced in-plane with respect to the ultrasound probe targeting the plane superficial to the serratus muscle. Under continuous ultrasound guidance a bolus of 30 ml of 0.25% levobupivacaine 30 min before skin incision. At the end of surgery, surgeon will put the catheter deep to serratus muscle and get it out with chest tube and fix it followed by an infusion of 5 ml/hour of 0.125% Levobupivacaine.
  Interventions: Procedure: Serratus anterior block

INTERVENTIONS:
Procedure: Serratus anterior block — after induction of anesthesia and Patients will be placed in the lateral position with the diseased side up. A linear ultrasound transducer (10-12 MHz) will be placed over the mid-axillary region of the thoracic cage in a sagittal plane. The rib will be counted inferiorly and laterally, until the fifth rib is identified in the mid-axillary line. The following muscles will be identified easily overlying the fifth rib: the latissimus dorsi (superficial and posterior), teres major (superior) and serratus muscle (deep and inferior). The needle (22- G, 50 - mm Touhy needle) will be introduced in-plane with respect to the ultrasound probe targeting the plane superficial to the serratus muscle. Under continuous ultrasound guidance a bolus of 30 ml of 0.25% levobupivacaine 30 mint before skin incision. At the end of surgery, surgeon will put the catheter deep to serratus muscle and get it out with chest tube and fix it followed by an infusion of 5 ml/hour of 0.125% Levobupivacaine.
  Arms: Serratus plane block
Procedure: thoracic epidural — In group I: thoracic epidural inserted at low thoracic level in sitting position then test dose will be administered to detect any complications then a bolus of 10 ml of 0.25% levobupivacaine 30 mint before skin incision followed by an infusion of 5 ml/hour of 0.125% levobupivacaine after surgery.
  Arms: Thoracic epidural

SUMMARY:
This study aims at comparing the effect of serratus plane block versus thoracic epidural in patients undergoing thoracotomy for lung cancer surgery regarding pain control and possible side effects.

DETAILED DESCRIPTION:
Introduction:

One of the most painful devastating surgical incisions is post-thoracotomy pain which can occur secondary to skin incision, damage to serratus anterior and intercostal muscles, rib retraction and injury of the intercostal nerves (1). It leads to pulmonary complications in the short term and chronic post-thoracotomy pain in the long term (2). The thoracic epidural is usually used as the reference analgesic approach for controlling thoracotomy pain (3) but it carries several risks and limitations (4). Serratus anterior plane block is performed by blocking the lateral cutaneous branches of the intercostal nerves (5) and can be a possible alternative to epidural block with lesser risks (6).

Aim of the work This study aims at comparing the effect of serratus plane block versus thoracic epidural in patients undergoing thoracotomy for lung cancer surgery regarding pain control and possible side effects.

Authors suggest that this technique is easy to perform, safe, effective with lesser side effects.

Study Design A randomized controlled study. Methodology

After approval of the institutional board ethical committee, written informed consent will be taken from the patients undergoing the study. Sixty patients between 20 to 60 years old undergoing thoracic surgery will be included in the study and randomly allocated into one of the two study groups:

Group (I) 30 patients: will receive 10 mL bolus of levobupivacaine 0.25% 30 mint before skin incision followed by an infusion of 5 ml/hour of 0.125% levobupivacaine after surgery.

Group (II) 30 patients: will receive 30 ml bolus of 0.25% levobupivacaine 30 mint before skin incision followed by an infusion of 5 ml/hour of 0.125% levobupivacaine after surgery.

Interventions:

Routine preoperative assessment will be conducted as standard (Complete blood count, liver, and kidney function tests, coagulation profile and chest x-ray) in addition to pulmonary function tests.

Upon arrival to the holding area, all the patients will be monitored by standard monitoring (ECG, Pulse oximetry and non-invasive automated arterial blood pressure). Then all patients will be pre-medicated with midazolam (3-5 mg intravenous) after fixation of 20 G cannula.

In group I: thoracic epidural inserted at a low thoracic level in sitting position then test dose will be administered to detect any complications, then a bolus of 10 ml of 0.25% levobupivacaine 30 mint before skin incision followed by an infusion of 5 ml/hour of 0.125% levobupivacaine after surgery.

In group II: after induction of anesthesia and Patients will be placed in the lateral position with the diseased side up. A linear ultrasound transducer (10-12 MHz) will be placed over the mid-axillary region of the thoracic cage in a sagittal plane. The rib will be counted inferiorly and laterally until the fifth rib is identified in the mid-axillary line. The following muscles will be identified easily overlying the fifth rib: the latissimus dorsi (superficial and posterior), teres major (superior) and serratus muscle (deep and inferior). The needle (22- G, 50 - mm Touhy needle) will be introduced in-plane with respect to the ultrasound probe targeting the plane superficial to the serratus muscle. Under continuous ultrasound guidance a bolus of 30 ml of 0.25% levobupivacaine 30 mint before skin incision. At the end of the surgery, the surgeon will put the catheter deep to serratus muscle and get it out with chest tube and fix it followed by an infusion of 5 ml/hour of 0.125% levobupivacaine.

Pain Management:

Intraoperative: by bolus dose for both groups. To ensure adequate analgesia throughout the operation all patients will be closely observed and upon the appearance of signs of inadequate analgesia e.g. increase in heart rate or systolic blood pressure 20% above the baseline, fentanyl rescue doses of 0.5µ/kg will be supplemented and recorded.

Postoperative: by continues infusion for both groups. All patients will have Intravenous paracetamol every 8 hours. Morphine 5mg intravenous will be given when the visual analogue scale (VAS) pain score becomes >3 as rescue analgesia.

Sample size:

The sample size was calculated based on the previous paper (7) estimating the difference in pain score at 24 h between 2 groups will be 2±2.1. Using power 80% and 5% significance level of 18 patients in each group will be sufficient to be able to reject the null hypothesis that the population means of the experimental and control groups are equal. This number is to be increased to 21 in each group to correct for non-parametric usage. Sample size calculation was achieved using Power and Sample Size Calculation Software Version 3.1.2 (Vanderbilt University, Nashville, Tennessee, USA).

Statistical analysis:

Data will be analyzed using Statistical Package for the Social Sciences (SPSS) win statistical package version 17. Parametric demographic data will be analyzed using student's t-test, Qualitative data will be compared using Chi-square test or Fisher's exact as appropriate. Numerical data will be described as mean and standard deviation (SD) or median and range as appropriate. While qualitative data will be described as frequency and percentage. P<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 60
* American Society of Anesthesiologists (ASA) physical status I-II grade
* Body mass index (BMI) < 40 kg/m2
* Undergoing elective thoracic surgery.

Exclusion Criteria:

* Coagulation defects
* Refusal for serratus anterior block
* Inability to obtain informed consent
* Local infection at the site of injection
* Bone metastases
* Known allergy to any of the used drug

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Score of postoperative pain at rest (Visual Analogue Scale, VAS, pain score). | 24 hours postoperative
  Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm)

SECONDARY OUTCOMES:
Score of postoperative pain at coughing (Visual Analogue Scale, VAS, pain score) | 24 hours postoperative
  Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm)
Amount of postoperative opioid consumption | 24 hours postoperative
No of patients developed adverse effects. | 24 hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute - Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP